CLINICAL TRIAL: NCT05227885
Title: The Effects of Nutritional Status and Habits on Disease Activity, Quality of Life and Functional Status of Patients in Rheumatoid Arthritis.
Brief Title: The Effects of Nutritional on Disease Activity and Functional Status in RA
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Bilal Uysal, Principal Investigator, Balikesir University
Other Study IDs: BalikesirUniversty
Record Dates: First submitted 2022-01-06; First posted 2022-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, nutrition, inflammation
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire form — A questionnaire will be applied to all participants. A questionnaire form will be applied to collect data on demographic information, pain, disease activity, nutritional habits, physical activity status and physical functional status of the patients included in the study.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic, autoimmune, systemic, inflammatory disease.

RA is a chronic inflammatory disease in which many patients cannot achieve remission despite current pharmacological treatments. Chronic inflammation in RA causes an increase in metabolic index and nutritional requirements. In recent studies, it is mentioned that diet regimens and foods consumed in nutrition affect inflammation.

The aim of this study is to evaluate the nutritional status and habits of patients with RA and to examine their effects on disease activity level, quality of life and functional status.

A questionnaire form will be applied to collect data on demographic information, disease activity, nutritional status and habits, physical activity status and physical functional status of the patients included in the study.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, autoimmune, systemic, inflammatory disease affecting 0.5-1.0% of the population. RA is a chronic inflammatory disease in which many patients cannot achieve remission despite current pharmacological treatments. Chronic inflammation in RA causes an increase in metabolic index and nutritional requirements. In recent studies, it is mentioned that diet regimens and foods consumed in nutrition affect inflammation.

The aim of this study is to evaluate the nutritional status and habits of patients with RA and to examine their effects on disease activity level, quality of life and functional status.

This study will be conducted with 100 patients diagnosed with RA in Balıkesir University, Health Practice and Research Hospital, Department of Physical Medicine and Rehabilitation outpatient clinic.

Patients between the ages of 18-75, diagnosed with RA according to the ACR 2010 diagnostic criteria, with a disease duration of 2 or more, using less than 10 mg of prednisolone per day, will be included in the study. Patients with a duration of ≤2 years after the diagnosis of RA, a change in the use of DMARDs and/or biological agents in their medical treatment for the last 8 weeks, using prednisolone more than 10 mg daily, malignancy, pregnant, lactating, and those who cannot understand the information in the questionnaire was not included in the study.

A questionnaire form will be applied to collect data on demographic information, disease activity, nutritional status and habits, physical activity and physical functional status of the patients included in the study.

As a result of this study, it is aimed to help patients with rheumatoid arthritis reach remission with diet programs and recommendations in addition to existing drug treatments.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75,
* Diagnosed with RA according to ACR 2010 diagnostic criteria,
* RA disease duration at least ≥2 years

Exclusion Criteria:

* Pregnant
* During the lactation period,
* Malignancy
* Using more than 10 mg of prednisolone per day,
* The period after the diagnosis of Ra is ≤2 years,
* Changes in medical treatment, DMARD and/or biological agent use in the last 8 weeks,
* Patients who cannot understand the information in the questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years, with a disease duration of at least 2 years or more, diagnosed with RA according to ACR 2010 diagnostic criteria,
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
A questionnaire form | Through study completion, an average of 4 month
  A questionnaire form to evaluate the demographic information
Nutritional status and habits; | Through study completion, an average of 4 month
  * Nutrient consumption frequencies
  * 24-hour retrospective food consumption record
Functional status of the patients. | Through study completion, an average of 4 month
  HAQ (Health Assessment Questionnaire)
Disease activity of the patients | Through study completion, an average of 4 month
  Simple Disease Activity Index (SDAI)

CONTACTS AND LOCATIONS:
Overall Officials: Bilal UYSAL, MD, Principal Investigator — Balikesir University
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided